CLINICAL TRIAL: NCT03384498
Title: Genetic Epidemiology of Malaria and Associated Antimalarial Drug Resistance
Brief Title: Malaria Genetic Surveillance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: BIOINF1602
Record Dates: First submitted 2016-08-18; First posted 2017-12-27 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Plasmodium Falciparum and Plasmodium Vivax
Keywords: Genetic epidemiology; Antimalarial drug resistance
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A fingerprick blood sample will be obtained to perform a malaria rapid diagnostic test or blood smear as part of standard care for malaria.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to determine the prevalence and geographical distribution of antimalarial drug resistance-linked genetic mutations in clinical P. falciparum and/or P.Vivax infection in the Greater Mekong Subregion

DETAILED DESCRIPTION:
This is a prospective observational study of patients with clinical Plasmodium falciparum and/or Plasmodium Viviax infection using parasite DNA from point-of-care fingerprick dried blood spot samples as well as a short survey on patient demographics, employment, travel, and mobile phone use to study P. falciparum parasite genotypes, population characteristics, and gene flow patterns.

On inclusion in the study and before standard treatment is administered, dried blood spots (DBS) will be obtained through fingerprick blood sampling from patients, with two or three blood spots on one piece of filter paper being obtained from each patient. Each blood spot will contain ~20µl of blood, for a total of ~ 40-60 uL of blood being collected from each patient for the study.

In order to have a greater understanding of the possible sites of malaria transmission and to relate genetic diversity to geographic location, patients or their parents/guardians will also be asked a short set of questions on demographics, their places of residence and work, recent mobile phone use, and their history of travel. The basic questions on phone utilisation will provide information on the use of mobile phones in the study population, including which mobile phone companies are used, and how many SIM cards and handsets each person carries. It will be employed to derive information on population movement from anonymised, aggregated data on mobile phone telephone use, i.e. call detail records (CDR), obtained from mobile phone companies in each country. This will be used for the modelling of population movement, its impact on the distribution of malaria and antimalarial drug resistance, and subsequent prediction of potential routes of spread of malaria and antimalarial drug resistance. As some of this information can be sensitive, during the consent process the patient will be given the option of not providing some or all of this information without needing to provide a reason. For those who do not wish to provide information, this will be documented in the survey form. A duplicate of the sample barcode will be placed on this same form, so the information therein can be matched with the relevant blood spot and its related genetic data, while retaining sample anonymity.

All patients in the study will receive standard care for falciparum malaria including drug therapy according to the national treatment guidelines of their country.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age
* P. falciparum and/or P.Vivax malaria as confirmed by positive rapid diagnostic test or asexual forms of P. falciparum on blood smear microscopy (may be mixed with non-falciparum Plasmodium species)
* Written informed consent by patient, parent/guardian, or legally authorised representative to participate in the study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages with P. falciparum and/or P.Vivax malaria who present to participating health facilities in Vietnam, Cambodia, Lao PDR, Thailand and Myanmar are the target study population.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Annual maps and reports on the prevalence of drug resistance-linked genetic mutations in P. falciparum parasites in the Greater Mekong Subregion | up to 12 months

SECONDARY OUTCOMES:
Allelic variations associated to drug resistance in P. falciparum at the locations surveyed | up to 12 months
  By using genotypes produced by high-throughput techniques (sequencing, PCR, mass spectrometry etc.).
Allelic variations associated to drug resistance in P. vivax at the locations surveyed | up to 12 months
  By using genotypes produced by high-throughput techniques (sequencing, PCR, mass spectrometry etc.).
Genetic differentiation between parasites populations at different locations in the Greater Mekong Subregion | up to 12 months
  By using population genetic measures such as FST and allele frequencies
Population structure of parasites | up to 12 months
  By using population genetics and clustering techniques, such as Principal Component Analysis and phylogeny
Gene flow patterns of P. falciparum malaria parasites in the Greater Mekong Subregion | up to 12 months
Likely geographic origin of P. falciparum malaria parasites in the Greater Mekong Subregion | up to 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- National Centre for Malaria Control, Parasitology and Entomology (CNM), Phnom Penh, Cambodia
- Center of Malariology, Parasitology and Entomology, Vientiane, Laos
- Institute of Malariology, Parasitology, and Entomology Quy Nhon, Qui Nhon, Vietnam

IPD SHARING:
Plan to Share IPD: Yes